CLINICAL TRIAL: NCT04911608
Title: Neuroendocrine Changes After Cervical Spinal Manipulation and Mobilization in Subjects With Non-specific Mechanical Neck Pain
Brief Title: Neuroendocrine Changes in Cervical Spinal Manipulation and Mobilization Non-specific Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Everett Lohman, Assistant Dean for Graduate Academic & Research Affairs Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5210211
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cervical manipulation (Experimental): The cervical spinal manipulation will consist of one session of a standard technique that will be performed by an experienced (>10 years) doctor of physical therapy practitioner. The technique is described by Gibbons and Tehan as a high-velocity, mid-range, low amplitude force at the segment of pain and/or segmental restrcition. The participant will lay comfortably in a supine position, the practitioner will then use his clinical discretion to select the most appropriate or symptomatic cervical motion segments and attempt to localize the manual thrust at those levels. A maximum of 2 attempts for each side of the cervical spine will be allowed regardless of the having achieved joint cavitation. This type of cervical manipulation procedure is described by Gibbons and Tehan as "Minimal Leverage Thrust" and it results in optimal patient comfort while receiving the treatment thus reducing post-treatment soreness/pain.
  Interventions: Other: cervical spinal manipulation
- cervical mobilization (Experimental): The cervical spinal mobilization treatment will also consist of one session of a standard technique that will be performed by an experienced (>10 years) doctor of physical therapy practitioner. For this procedure, the participant will lay comfortably in a prone position, the practitioner will then use his clinical discretion to select the most appropriate or symptomatic cervical motion segments and attempt to localize the manual forces at those segments. The magnitude of a mobilization-or how hard the therapist pushes on the spine-is usually reported as the magnitude of force. For an oscillatory posterior-anterior (PA) mobilization technique, the maximum magnitude of applied force is usually reported as the mean of the force peaks that occur during a specified period.34 The cervical mobilization will consist of oscillations of 1Hz and magnitude forces of 30 Newtons (N) for 30 seconds, 90N for 120 seconds and 30N for 30 seconds at the localized segment.
  Interventions: Other: cervical spinal mobilization
- postural correction education (No Intervention): Participants will be presented with a standardized educational short video regarding the importance of postural correction movements.

INTERVENTIONS:
Other: cervical spinal manipulation — High-velocity, mid-range, low amplitude force at the segment of pain and/or segmental restriction. The participant will lay comfortably in a supine position, the practitioner will then use his clinical discretion to select the most appropriate or symptomatic cervical motion segments and attempt to localize the manual thrust at those levels. A maximum of 2 attempts for each side of the cervical spine will be allowed regardless of the having achieved joint cavitation.
  Arms: cervical manipulation
Other: cervical spinal mobilization — Participant will lay comfortably in a prone position, the practitioner will then use his clinical discretion to select the most appropriate or symptomatic cervical motion segments and attempt to localize the manual forces at those segments.
  Arms: cervical mobilization

SUMMARY:
The aim for this graduate student research project is to determine if cervical spinal mobilization releases similar neuropeptides and endogenous hormones as compared to cervical spinal manipulation and a control group. We hypothesized that application of cervical manipulations would result in a neuroendocrine response (SNS- HPA axis). By measuring salivary cortisol, oxytocin and DHEA, it may be possible to provide important information regarding the mechanisms and associations of pain modulation, anti-inflammatory and tissue healing after a biomechanical event.

DETAILED DESCRIPTION:
* Participants will be completing three standardized questionnaires: The Neck Disability Index (NDI), Numeric Pain Rate Scale (NPRS), and the Global Ration of Change (GROC). These self-rated questionnaires will be used to capture the patient's level of pain, assess disability, and to quantify patient's improvement or deterioration over time, usually to either determine the effect of an intervention or to chart the clinical course of a condition.
* Participants will be providing four saliva samples: Collecting biomarkers in saliva requires reliable, accurate methods for proper storage and handling techniques with high-quality assays and validated testing protocols. For this study, salivary oxytocin, cortisol and dehydroepiandrosterone (DHEA) will be collected in the morning (between 8 am and 11 am) for each participant at preintervention (baseline), and 15, 30 and 60 minutes after intervention by using self-collection kits in accordance with the manufacturer's instructions for each biomarker (Salimetrics Inc).
* Participants will be receiving skilled interventions: Participants will be randomly assigned by using a computer-generated randomized table of numbers created prior to the start of data collection to one of the following three groups: cervical manipulation group, cervical mobilization group, no-touch group which will be receiving postural education. Cervical Spinal Manipulation (CSM) and Cervical Spinal Mobilizations (CSMob) are common techniques utilized by healthcare professionals to treat neck pain, low back pain and its effectiveness to treat musculoskeletal pain.

ELIGIBILITY:
Inclusion Criteria:

1. . Subjects will be healthy male and females between 18 to 60 years of age.
2. . Resting neck pain ≤ 30 days that is mechanical in nature without radiating pain below shoulder.
3. . Neck Disability Index ≥ 10/50.
4. . Negative Upper Cervical instability tests such as Sharper-Purser test, Alar ligament test and Transverse ligament test.

Exclusion Criteria:

1. . Cervical Arterial Dysfunctions.
2. . Serious medical conditions (CA, spinal cord injury).
3. . History of instability disorders (History of neck injury, surgery, fractures, osteoporosis, arthritis, ankylosing spondylitis).
4. . Neurological conditions (Nerve root compression, central nervous system involvement, myelopathy, fibromyalgia.
5. . Endocrine dysfunctions (Autoimmune-related diseases, adrenal gland pathology, systematic metabolic disorders).
6. . Pregnancy/Lactating/Postpartum.
7. . Pending legal action regarding their neck pain.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | change between baseline and 2 days
  Survey used to assess self-rated disability in patients with neck pain.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | change between baseline and 2 days
  The questionnaire is used to capture the patient's level of pain by using an 11-point scale, ranging from 0 (no pain) to 10 (worst pain imaginable).
Global Ratio of Change | change between baseline and 2 days
  This is a 15-point scale to rate the patient's own perception of improved or deteriorated function.
Salivary Biomarkers | change between baseline and 15, 30 and 60 minutes after intervention.
  Salivary oxytocin, cortisol and dehydroepiandrosterone (DHEA) will be collected for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Everett Lohman, Dsc, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States